CLINICAL TRIAL: NCT04968834
Title: Protocol For Genomically Profiling, Collecting, Archiving And Distributing Blood And Bone Marrow Specimens From Children And Young Adults With Hematologic Malignancy
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Charles H. Hood Foundation (Other); Rally Foundation for Childhood Cancer Research (Other)
Responsible Party: Principal Investigator, Yana Pikman, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 20-302
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myeloproliferative Syndrome
Keywords: Leukemia; Myelodysplastic Syndromes; Myeloproliferative syndrome (MPS)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Genetic Profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOMIC PROFILING AND SPECIMEN BANKING REGISTRATION ARM: The research study procedures include screening for eligibility, reviewing and signing this consent form, collecting patient information and clinical data, obtaining previously collected bone marrow and blood samples, and completing a brief optional Household Survey. Bone marrow and blood samples may also be collected in the future as part of your routine clinical procedures
  Interventions: Genetic: Genomic profiling

INTERVENTIONS:
Genetic: Genomic profiling — Genomic profiling using CLIA assay

SUMMARY:
This research study is a genomic profiling and repository study for children and young adults who have leukemia, myelodysplastic syndrome (MDS) or myeloproliferative syndrome (MPS). Genes are the part of cells that contain the instructions which tell cells how to make the right proteins to grow and work. Genes are composed of DNA letters that spell out these instructions. Genomic profiling helps investigators understand why the disease develops and the instructions that led to its development. Understanding the genetic factors of the disease can also help investigator understand why the disease of some people can respond to certain therapies differently than others.

The genomic profiling will be performed using bone marrow and blood samples that either have already been obtained during a previous clinical procedure or will be obtained at the time of a scheduled clinical procedure. Studying the genetic information in the cells of these samples will provide information about the origin, progression, and treatment of leukemia and myeloproliferative syndromes and myelodysplastic syndrome. Storing the bone marrow and blood samples will allow for additional research and genomic assessments to be performed in the future.

DETAILED DESCRIPTION:
Pediatric patients with new diagnosis or relapsed/refractory acute leukemia, MDS/AML, chronic leukemia, myeloproliferative syndromes or myelodysplastic syndrome will be enrolled onto this study. At the time of enrollment, a sample of the leukemia will be submitted for genomic profiling using CLIA assay(s). This information will be returned to the treating oncologist. The study will collect follow up data on patient outcome and whether the genomic profiling influenced treatment.

It is expected that about 100 people each year will take part in this research study at 8 medical centers in the United States

ELIGIBILITY:
Inclusion Criteria:

* Age: birth to < 30 years of age
* Diagnosis:

  -- Patient with acute leukemia, chronic leukemia, MDS/AML, myelodysplastic syndrome or myeloproliferative syndromes. Disease can be newly diagnosed or relapsed/refractory.
* Pathology Criteria:

  -- Histologic confirmation of leukemia or myelodysplastic syndrome (MDS) or myeloproliferative syndrome (MPS) at the time of diagnosis or recurrence
* Specimen Criteria:

  * Sufficient sample available for genomic profiling OR bone marrow aspirate/blood draw planned for clinical care which is anticipated to allow collection of minimum specimen for testing (See Section 6.1 for description of specimen requirements)

Exclusion Criteria:

- Insufficient leukemia or MDS specimen available for profiling from diagnosis or recurrence (See Section 6.1); or bone marrow evaluations NOT planned for clinical care; or peripheral blast percentage <20%, or clinical blood draw not planned

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - birth to < 30 years of age. Patient with acute leukemia, chronic leukemia, MDS/AML, myelodysplastic syndrome or myeloproliferative syndromes. Disease can be newly diagnosed or relapsed/refractory.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Enrolled for Genomic Profiling-Pediatric Leukemia | 3 Years
  To perform genomic profiling of pediatric leukemia using clinical genomics platforms and return results to treating oncologist. This objective will be accomplished by enrolling patients and obtaining samples for sequencing and banking. The pathologist-interpreted genomic test results will be returned to the treating oncologist.

SECONDARY OUTCOMES:
Number of Patients Enrolled for Genomic Profiling-New Diagnosis | 3 Years
  To collect and bank samples from pediatric patients with new diagnosis or relapsed/refractory acute and chronic leukemia, and myelodysplastic syndrome. This objective will be accomplished by enrolling patients and obtaining samples for sequencing and banking.

CONTACTS AND LOCATIONS:
Overall Officials: Yana Pikman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Maine Medical Center, Portland, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Lifespan Cancer Institute, Providence, Rhode Island
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu